CLINICAL TRIAL: NCT02161445
Title: Systolic Time Intervals: a Diagnostic Tool of Acute Heart Failure in Emergency Departement Settings
Brief Title: Systolic Time Intervals in the Diagnosis of Heart Failure in Emergency Departement
Acronym: STA/AHF
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: STI in AHF
Record Dates: First submitted 2014-05-04; First posted 2014-06-11 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Dyspnea
Keywords: impedance; pep; tevg; dyspnea; AHF; BNP
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AHF group: patients with AHF diagnosed based on clinical, biological and echocardiographic findings. Two sub-groups of patients were identified within HF group: Patients with reduced (<45%) LVEF (HFrEF) and those with preserved (≥45%) LVEF (HFpEF).
  Interventions: Device: the acoustic cardiographic parameters were calculated
- non AHF group: we included patients with acute dyspnea and for whom acute heart failure was excluded
  Interventions: Device: the acoustic cardiographic parameters were calculated

INTERVENTIONS:
Device: the acoustic cardiographic parameters were calculated — STIs were measured using simultaneous recording of the electrocardiogram and acoustic cardiography signals using an analogic numeric system (Biopac Systems, Goleta, CA). A3-minute acoustic cardiographic tracing for all patients was obtained and stored electronically. We measured the electromechanical activation time (EMAT) which is the time between the initial deflection of the electrocardiographic Q wave and the first phonocardiographic complex corresponding to the first heart sound (S1). The left ventricle ejection time (LVET) defined as the interval between the peak components from the S1 and S2 complexes was measured on the same cardiac cycles. All studies were performed in patients in a semi-recumbent position with head at 30 degrees position. For each patient, the acoustic cardiographic parameters were calculated from a 10-second free of artifact recording of data averaging 8 to 12 beats measurements.

SUMMARY:
the gold standard for the diagnostic of acute heart failure is based on clinical, biological (BNP levels) and echocardiographic findings, but still in some cases, the diagnosis is difficult and requires further investigations.

BNP dosages and echocardiography are not always available in many medical centers, especially in emergency departements, and are expensive.

we investigated the use of alternative methods, such as the systolic time intervals (STI), in the diagnosis of acute heart failure (AHF) in emergency departement patients consulting for dyspnea.

DETAILED DESCRIPTION:
AHF is a common cause for dyspnea, but still hard to diagnose. in emergency departements, physicians dispose of a variety of techniques helping them to identify patients with acute onset dyspnea due to cardiac causes and allowing them to initiate the appropriate therapeutics.

techniques such as the N type brain natriuretic peptid (NT BNP) dosages and echocardiography, in addition to the clinical exam, are efficient in these cases but they encounter many problems:

* the BNP dosages are non-conclusive in some cases (grey zone) and must be repeated wich takes time.
* echocardiography is operator - dependent technique and could be misleading in some conditions.
* both BNP and echocardiography are expensive and not found in many emergency structures, especially in poor countries.

all the arguments pushed us to investigate other simpler and cheaper techniques to apply in these conditions.

STI is an old technique based on the recording of two parameters: electrocardiogram and phonocardiogram, and from them measuring the different systolic intervals:

* pre-ejection period (PEP): defined as the interval between the beginning of the QRS wave and the first heart sound (B1).
* electro-mechanic activation time (EMAT): defined as the interval between the two heart sounds B1 and B2
* the PEP / EMAT time in acute onset heart failure, the conduction times are increased, due to tissular lesions, which prolong the PEP, also the myocardial contractility is deficient and the heart puts less time to eject the blood volume which decrease the EMAT and in summary the PEP/EMAT is increased significatively.

in this study protocol, we aimed to investigate the diagnostic performance of STI compared to conventional methods in the diagnosis of acute heart failure in emergency department settings.

ELIGIBILITY:
Inclusion Criteria:

* non traumatic dyspnea
* age more than 18 years old.

Exclusion Criteria:

* ECG diagnostic for acute myocardial infarction or ischemic chest pain within the prior 24 hours
* history of a heart transplant
* pericardial effusion
* chest wall deformity suspected of causing dyspnea
* coma, shock,Mechanical Ventilation, vasopressor drugs
* arrhythmia serious and sustained, pace maker severe mitral valve disease, severe pulmonary arterial hypertension
* renal failure with creatinine >350micromol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged more than 18 years old presenting at the ED with non traumatic dyspnea.
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2012-10-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PEP/EMAT values between the AHF and non AHF groups | at admission (an average of 24 hours)
  compare the PEP/EMAT values between the two study groups: AHF and non-AHF. the diagnosis of AHF is made based on clinical, BNP, and echocardiographic findings.

SECONDARY OUTCOMES:
PEP values between the two study groups | at admission (an average of 24 hours)
  compare the PEP values between the two study groups: AHF and non-AHF. the diagnosis of AHF is made based on clinical, BNP, and echocardiographic findings.
compare the EMAT values between the two study groups | at admission (an average of 24 hours)
  compare the EMAT values between the two study groups: AHF and non-AHF. the diagnosis of AHF is made based on clinical, BNP, and echocardiographic findings.
compare the STI diagnostic performance against BNP | at hospital admission (an average of 24 hours)
  compare the diagnostic performance, based on the area under curve estimation of the ROC curve, between the STI (PEP, EMAT and PEP/EMAT) and the BNP levels

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Professor, Principal Investigator — University hospital of Monastir
Locations (1):
- Nouira Semir, Monastir, Emergency Department Monastir, Tunisia 5000, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com